CLINICAL TRIAL: NCT04098848
Title: The Effect of Intradialytic Exercise on the Fatigue, Sleep Disorder, Arterial Stiffness and Endothelial Function in Uremic Patients
Brief Title: Intradialytic Exercise on the Fatigue, Sleep Disorder, Arterial Stiffness and Endothelial Function in Uremic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB106-139-A
Record Dates: First submitted 2019-09-15; First posted 2019-09-23 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Hemolysis; Exercise; Sleep Disorder; Fatigue; Adipocytes
MeSH Terms: conditions — Hemolysis; Motor Activity; Sleep Wake Disorders; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradialytic exercise (Experimental): Cycling exercise 30 minutes a time, three times a week during hemodialysis
  Interventions: Other: Cycling exercise
- Control group (No Intervention): not participate in cycling exercise during hemodialysis

INTERVENTIONS:
Other: Cycling exercise — Intradialytic cycling exercise for 30 minutes a time
  Arms: Intradialytic exercise

SUMMARY:
To determine the effect of intradialytic cycling exercise on fatigability, sleep disorders, arterial stiffness and endothelial function in dialysis patients

DETAILED DESCRIPTION:
The endothelium is a key regulator of vascular homeostasis and chronic exposure to vascular risk factors alters the regulatory properties of the endothelium, which progresses toward a pro-inflammatory pattern, senescence, and apoptosis. Endothelial cell integrity and function are critical to the prevention of atherosclerosis, and therefore endothelial cell injury and dysfunction are major steps in the development and progression of cardiovascular disease. Endothelial dysfunction may be the landmark of active disease process through the course of atherosclerotic cardiovascular disease, and a significant risk factor for future cardiovascular events.

Several studies had reported that not only medical treatment but also exercise could improve physical and vascular functions, dialytic efficiency, quality of sleep, fatigue and depression et al. Exercise could be classified to aerobic, Anaerobic exercise and resistance et. Several studies have shown that regular cycling exercise in hemodialysis patients could improve physical activity, sleep quality, and reduce fatigability. Therefore, exercise plays an important role in hemodialysis patients. According to these benefits, the investigator's study was designed to explore the effects of intradialytic cycling exercise on sleep quality and fatigability, adipokines and myokinins levels in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Regular hemodialysis more than 3 months with 4 hours a time, thrice a week
* Eligible to sign permit

Exclusion Criteria:

* Could not sign permit or do not want to join the trial
* Infection
* Amputation of any one of the lower limb
* Hemodynamic unstable
* Acute myocardial infarction (AMI) in recent 6 months
* Unstable heart condition, such as unstable angina, arrythmia
* Deep vein thrombosis (DVT)
* History of kidney transplantation
* Vascular access over lower limb

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change of the Functional Assessment of Chronic Illness Therapy -Fatigue (FACIT-F) score for 2 years | pre-test and then every 3 months for 2 years
  Compare the FACIT-F score before, during and after intradialytic cycling exercise FACIT-F score is from 0-52 points; higher score represents less fatigue.
Change of the Pittsburgh Sleep Quality Index (PSQI) score for 2 years | pre-test and then every 3 months for 2 years
  Compare the PSQI score before, during and after intradialytic cycling exercise PSQI score is from 0-21 points; score>=5 means poor sleeping quality.
Change of the carotid-femoral pulse wave velocity (cfPWV) for 2 years | pre-test and then every 3 months for 2 years
  Compare the cfPWV before, during and after intradialytic cycling exercise
  cfPWV measurement: a measure of aortic wall stiffness, increases markedly with age. Each set of pulse wave and ECG data to calculate the mean time difference between R-wave and pulse wave on a beat-to-beat basis, with an average of 10 consecutive cardiac cycles. The cfPWV will be calculated using the distance and mean time difference between the two recorded points.
  Patients with cfPWV values of > 10 m/s were classified in the high arterial stiffness group, whereas those with cfPWV values of ≤10 m/s were assigned to the low arterial stiffness group.
Change of the cardio-ankle vascular index (CAVI) for 2 years | pre-test and then every 3 months for 2 years
  Compare the CAVI before, during and after intradialytic cycling exercise
  CAVI is a novel and accurate method, independent of the effect of blood pressure, and is used as a predictor of arterial stiffness (AS) AS was defined as a CAVI ≥ 9
Change of the brachial-ankle pulse wave velocity (baPWV) for 2 years | pre-test and then every 3 months for 2 years
  Compare the baPWV before, during and after intradialytic cycling exercise
  baPWV is one measure arterial stiffness using brachial to ankle arterial wave analyses and has been used to assess peripheral arterial stiffness (PAS)
  baPWV value >14.0 m/s on either side was considered high PAS.
Change of the aortic augmentation index(AI) measurements for 2 years | pre-test and then every 3 months for 2 years
  Compare the AI before, during and after intradialytic cycling exercise
  AI of central blood pressure have been widely used as clinical indices of arterial stiffness AI is an indirect measure of central arterial stiffness, but mainly a direct measure of central wave reflection
Change of the brachial flow-mediated vasodilatation (bFMD) for 2 years | pre-test and then every 3 months for 2 years
  Compare the bFMD before, during and after intradialytic cycling exercise
  Endothelial function is often quantified by FMD, which represents the endothelium-dependent relaxation of a conduit artery-typically the brachial artery - due to an increased blood flow.
Change of the digital thermal monitoring (DTM) for 2 years | pre-test and then every 3 months for 2 years
  Compare the DTM before, during and after intradialytic cycling exercise
  DTM is a simple noninvasive method to measure endothelial function and vascular reactivity that is correlated with atherosclerosis risk factors and coronary artery disease
  Vascular reactivity index (VRI) < 1.0: the poor vascular reactivity, 1.0 ≤ VRI < 2.0: the intermediate vascular reactivity, and VRI ≥ 2.0: the good vascular reactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsien Lai, Principal Investigator — Attending physician
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No